CLINICAL TRIAL: NCT01467765
Title: The Comparative Study of Elemental Diet and Regular Liquid Diet on Gastric Emptying in Patients With Percutaneous Endoscopic Gastrostomy
Brief Title: The Effect of Elemental Diet on Gastric Emptying
Acronym: Elental
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Digestive Disease Center, Showa Inan General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Elental study
Record Dates: First submitted 2011-11-05; First posted 2011-11-09 (Estimated); Last update posted 2012-08-09 (Estimated); Status verified 2012-08

CONDITIONS: Postprocedural Delayed Gastric Emptying

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elemental diet (Active Comparator)
  Interventions: Other: Elental
- Liquid nutrient (Placebo Comparator)
  Interventions: Other: Elental

INTERVENTIONS:
Other: Elental — 200Kcal/200mL of liquid nutrient for 15 min at 7:30 am is administered in PEG patients

SUMMARY:
In patients with percutaneous endoscopic gastrostomy (PEG) delayed gastric emptying has been speculated as a cause of aspiration pneumonia. Elemental diet may facilitate gastric emptying in PEG patients as compared with regular liquid enteral nutrients, resulting in the prevention of aspiration pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* percutaneous endoscopic gastrostomy patients

Exclusion Criteria:

* history of abdominal surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Measurement of gastric emptying | Four hours (from 7:30 am to 11:30 am)
  Two kinds of liquid test meals (Elemenal diet or regular liquid nutrient ) (200kcal/200ml) labeled with 100 mg(13C sodium acetate) are administered for 15 min and after that 13C breath test performed during the 4 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Showa Inan General Hospital, Komagane, Nagano, Japan